CLINICAL TRIAL: NCT03071146
Title: A Prospective Study of the Performance of the Bard LifeStent 5F Vascular Stent System
Brief Title: Utility, Safety, and Effectiveness of the Bard LifeStent 5F Vascular Stent System
Acronym: REALITY III
Status: Completed | Type: Observational
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Other Study IDs: BPV-16-004
Record Dates: First submitted 2017-02-21; First posted 2017-03-06 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Peripheral Arterial Disease; Intermittent Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bard® LifeStent® 5F Vascular Stent System: Patients with lesion(s) in the infra-inguinal segment (SFA and/or popliteal artery) will be treated with percutaneous transluminal angioplasty (PTA) and the Bard® LifeStent® 5F Vascular Stent System.
  Interventions: Device: Bard® LifeStent® 5F Vascular Stent System

INTERVENTIONS:
Device: Bard® LifeStent® 5F Vascular Stent System — The LifeStent® Vascular Stent is a peripheral stent intended to improve luminal diameter in the treatment of symptomatic de-novo or restenotic lesions up to 240 mm in length in the native superficial femoral artery (SFA) and popliteal artery with reference vessel diameters ranging from 4.0 - 6.5 mm.

SUMMARY:
The medical device being examined in this study is the Bard® LifeStent® 5F Vascular Stent System. It is intended for use in patients who suffer from peripheral artery disease (PAD). PAD is generally associated with blocked arteries of the legs. The superficial femoral artery (SFA) and popliteal artery are common locations for this problem to develop. The patient may experience pain or discomfort in the leg that occurs when walking or have other complications associated with wound healing. The purpose of this study is to collect information to assess the deliverability, clinical utility, safety and effectiveness of the Bard® LifeStent® 5F Vascular Stent System.

ELIGIBILITY:
Inclusion Criteria:

* The subject or legal representative has been informed of the nature of the evaluation, agrees to its provisions, and has signed the informed consent form (ICF).
* Subject agrees to comply with the protocol-mandated follow-up procedures and visits.
* The subject is ≥ 21 years of age.
* The subject has lifestyle-limiting claudication to mild tissue loss defined as: Rutherford Category 2-5 (moderate claudication to minor tissue loss).
* The target lesion(s) has angiographic evidence of a hemodynamically relevant stenosis or restenosis ≥50% or occlusion of the SFA and/or popliteal artery (by visual estimate) and is amenable to PTA and stenting.
* The target vessel reference diameter will be (by visual estimate) appropriate for treatment with available stent diameters of 5.0, 6.0 and 7.0 mm.
* A total of two stents may be used to treat a target lesion. Overlapping is allowed.
* There is angiographic evidence of at least one vessel runoff to the foot (at the level of the malleolus).

Exclusion Criteria:

* The subject is unable or unwilling to provide informed consent or is unable or unwilling to comply with the study follow-up procedure and visits.
* The subject has claudication or critical limb ischemia described as Rutherford Category 0 (asymptomatic), 1 (mild claudication), or 6 (major tissue loss).
* The subject has a known contraindication (including allergic reaction) or sensitivity to nickel, titanium or tantalum.
* The subject has a known allergy of hypersensitivity to contrast media which cannot be adequately pre-medicated.
* The subject has a known uncontrolled blood coagulation/bleeding disorder.
* The subject has concomitant renal failure with a creatinine of >2.5 mg/dL.
* The subject has concomitant hepatic insufficiency, thrombophlebitis, uremia, systemic lupus erythematosus (SLE), or deep vein thrombosis (DVT) at the time of the study procedure.
* The subject is receiving dialysis or immunosuppressive therapy.
* The subject is diagnosed with septicemia at the time of the study procedure.
* The subject is participating in an investigational drug or another investigational device study.
* The subject has another medical condition, which, in the opinion of the investigator, may cause him/her to be noncompliant with the protocol, confound the data interpretation, or is associated with limited life expectancy not sufficient to complete all study procedures.
* The subject has extensive peripheral vascular disease, which, in the opinion of the investigator, precludes safe insertion of an introducer sheath.
* The target lesion is located within an aneurysm or associated with an aneurysm in the vessel segment either proximal or distal to the target lesion.
* The subject has angiographic evidence of poor inflow, which would be deemed inadequate to support a vascular bypass graft.
* The subject has severe calcification of the target lesion, which prevents inflation of a PTA balloon (pre-dilatation of the target lesion is required).
* The subject has angiographic evidence of large acute thrombus at the target lesion.
* Subjects with a stent previously implanted into the target lesion. A target vessel with a previously placed stent is permitted as long as the subject device(s) will not come into contact with the previously placed stent during treatment of the target lesion.
* Lesion requiring the use of more than two stents.
* Bilateral disease in the native SFA and/or popliteal artery where both limbs meet the inclusion/exclusion criteria and it is planned to treat both limbs within 30 days. Note: One limb may be enrolled in the study, but only if the second limb is planned to be treated after the 30 day follow-up telephone screening has taken place. The limb that may be enrolled has to be the limb with the more severe lesion and the reasons for treating this specific limb will need to be stated in the case report form (CRF).
* The subject had a prior vascular intervention within 30 days before, or has an intervention planned for within 30 days after the index procedure. Note: Additional non-target lesions may be treated during the index procedure.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted among patients who are candidates for PTA and stenting with lesion(s) in the infra-inguinal segment (SFA and/or popliteal artery).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Freedom from occurrence of death | 30 days post-index procedure
Freedom from occurrence of amputation | 30 days post-index procedure
Freedom from TLR (Target Lesion Revascularization) | 30 days post-index procedure
  TLR is defined as a revascularization procedure (e.g. PTA, cryoplasty, etc.) of the target lesion.
Freedom from TVR (Target Vessel Revascularization) | 30 days post-index procedure
  TVR is defined as a revascularization procedure (e.g. PTA, stenting, surgical bypass, etc.) of the target vessel outside the target lesion.
Technical success | At the time of index procedure (usually within 10 minutes)
  Technical success is defined as successful deployment and placement accuracy based upon a rating scale completed by the investigators. bookend sizes will be evaluated for clinical utility of size range.

SECONDARY OUTCOMES:
Freedom from TLR (Target Lesion Revascularization) | Up to 12 months post-index procedure
  TLR is defined as a revascularization procedure (e.g. PTA, cryoplasty, etc.) of the target lesion.
Freedom from TVR (Target Vessel Revascularization) | Up to 12 months post-index procedure
  TVR is defined as a revascularization procedure (e.g. PTA, stenting, surgical bypass, etc.) of the target vessel outside the target lesion.
Primary patency rates | Up to 12 months post-index procedure
  Patency is defined as a reduction in luminal diameter (stenosis) of <=50% and of <=70% measured by Duplex ultrasound (DUS) (peak systolic velocity ratio or PSVR <= 2.4 and <=3.4). Failure of primary patency is defined as a restenosis (reduction in luminal diameter of >50%) as measured by DUS (PSVR >2.4).
Freedom from death | 12 months post-index procedure
  TLR is defined as a revascularization procedure (e.g. PTA, cryoplasty, etc.) of the target lesion. TVR is defined as a revascularization procedure (e.g. PTA, stenting, surgical bypass, etc.) of the target vessel outside the target lesion.
Freedom from occurrence of stroke | 12 months post-index procedure
Freedom from occurrence of MI (myocardial infarction) | 12 months post-index procedure
Occurrence of emergent surgical revascularization of the target limb | 12 months post-index procedure
Occurrence of significant distal embolization in target limb | 12 months post-index procedure
Occurrence of target limb major amputation | 12 months post-index procedure
Occurrence of thrombosis of target vessel | 12 months post-index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zeller, MD, Principal Investigator — Universitaets-Herzzentrum Freiburg, Bad Krozingen
Locations (4):
- Germany (4):
  - Fuerst-Stirum-Klinik Bruchsal, Bruchsal, Gutleutstr. 1-14
  - Gemeinschaftspraxis fuer Radiologie, Berlin, Heinz-Galinski-Str. 1
  - Praxis fuer Interventionelle Angiologie, Kaiserslautern, Strassburger Allee 4
  - Universitaets-Herzzentrum Freiburg, Klinik fuer Kardiologie und Angiologie II, Bad Krozingen, Suedring 15

IPD SHARING:
Plan to Share IPD: No